CLINICAL TRIAL: NCT06086106
Title: Comparison Between the Caudal Block and Other Methods of Postoperative Pain Relief in Children Undergoing Circumcision: A Prospective Randomized Study"
Brief Title: Comparison Between the Caudal Block and Other Methods of Postoperative Pain Relief in Children Undergoing Circumcision
Acronym: paincontrol
Status: Completed | Type: Observational
Sponsor: Salmaniya Medical Complex (Other Government)
Responsible Party: Principal Investigator, Zeana gawe, Specialist Of Anesthesia, Salmaniya Medical Complex
Other Study IDs: 70130623
Record Dates: First submitted 2023-08-30; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Analgesia; Pain, Postoperative; Pain, Acute
Keywords: Anesthesia; Pain Management; pediatric
MeSH Terms: conditions — Agnosia; Pain, Postoperative; Acute Pain | interventions — Analgesics, Opioid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group B systemic opioids for pain relive: systemic opioids belong to a class of analgesics, they act by attaching to opioid receptors in the brain and spinal cord. For relief of pain, they are frequently utilized in a variety of surgical procedures and can be given intravenously, and in intramuscular injections. Although opioids are considered highly effective in pain control, they can lead to several adverse effects, such as nausea, vertigo, and respiratory depression, some of which can be dangerous.
  Interventions: Procedure: caudal block; Procedure: Dorsal Penile Nerve Block DPNB; Drug: Systemic opioids

INTERVENTIONS:
Procedure: caudal block — The caudal block involves the injection of a local anesthetic Bupivacaine dose of 0.75 to 1 ml/kg the maximum volume was 10 mL with 0.25% concentration into the caudal epidural space, targeting the sacral nerve roots. to provide a high effect and duration of analgesia
  Other Names: Regional anesthesia intervention
Procedure: Dorsal Penile Nerve Block DPNB — DPNB is A type of pain control post-operative, often performed as a circumferential infiltration of the root of the penis (ring block). Two skin wheals are raised at the dorsal base of the penis, one on each side just below and medial to the pubic spine. A 25-gauge, 37.5-mm needle is introduced on each side, and the bupivacaine (1 to 1.5 mL) maximum dose 2 ml concentration 0.25% for infants is injected superficially and deep along the lower border of the pubic ramus to anesthetize the dorsal nerve. For a complete ring of infiltration,
  Other Names: Regional anesthesia intervention.
Drug: Systemic opioids — Systemic opioids belong to a class of analgesics, they act by attaching to opioid receptors in the brain and spinal cord. For relief of pain, they are frequently utilized in a variety of surgical procedures and can be given intravenously, and in intramuscular injections. Although opioids are considered highly effective in pain control, they can lead to several adverse effects, such as nausea, vertigo, and respiratory depression, some of which can be dangerous.
  Other Names: opioids analgesic

SUMMARY:
Prospective, randomized, case-controlled trial study. Observation post-operatively:

Aims: This study aimed to compare the effectiveness of the caudal block CB with other methods of postoperative pain release.

DETAILED DESCRIPTION:
a study Sample size: all patients, for a total of 90 boys going for circumcision surgery. I was recruited over the course of four months, starting on 1 May 2023. The patients will be divided into three groups: A caudal block(CB), B systemic opioids, and C dorsal penile block (DPNB) Techniques used in pediatric surgeries to provide analgesia for penile surgery such as circumcision. All patients had operations and were observed, and the three groups were compared based on hemodynamic stability, pain scores, duration of sedation, analgesia need, and parental satisfaction. where the Face, Leg, Activity, and Cry Consolability (FLACC) pain scale and behaviors were used to observe and compare the three groups. Pain scores were recorded by separate anesthesiologists or nurses in the post-anesthesia care unit. All statistical work will be carried out using Spss version 27 (Spss Inc., Chicago, USA) and Prism GraphPad version 9.4.1 (GraphPad, San Diego, USA) The categorical and numerical variables and demographic data of three groups were collected and reviewed by two authors. the study has shown that the caudal block produces higher levels of analgesia and a longer period of pain release than the penile block, even if both methods help relieve pain during pediatric surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status classification one
* aged from three months up to three years

Exclusion Criteria:

* allergic to local anesthetics,
* bleeding diatheses,
* coagulopathy,
* infection at the injection site,

Ages: 3 Months to 3 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — patients, for a total of 90 boys going for circumcision surgery, aged from 3 months up to 3 years
Study Population: Prospective, randomized, case-controlled trial study. Observation post-operatively: a study Sample size: all patients, for a total of 90 boys going for circumcision surgery. I was recruited over the course of four months, starting in May 2023. The patients will be divided into three groups: A (CB), B systemic opioids, and C (DPNB). All patients had operations and were observed, and the three groups were compared based on hemodynamic stability, pain scores, duration of sedation, analgesia need, and parental satisfaction. where the Face, Leg, Activity, and Cry Consolability (FLACC) pain scale and behaviors were used to observe and compare the three
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
postoperative pain assessment | "immediately after the intervention/procedure/surgery"
  The circumcision of children is the most commonly performed surgical procedure in the world Likely, the greatest target for us as anesthesiologists is to control the pain postoperatively. Various techniques are used to manage pain. Two of these techniques are CB and DPNB, both considered as regional blocks and involve the administration of local anesthesia. Additionally, systemic opioids have shown potential for alleviating postoperative pain. This study aimed to explore the benefits and limitations of these techniques and provide insights into their effectiveness and impact on circumcised patients. By evaluating the use of CB, penile block, and opioids, we can recognize their usefulness in promoting safe and painless circumcision surgery.Considering the risk points, DPNB can cause hematoma, opioids can lead to respiratory depression plus nausea and vomiting, while CB can cause delayed micturition, failed block, and cerebrospinal fluid aspiration due to puncture of dura
Pain postoperative assessment tools in post anesthesia care unit. | 20 minutes after the intervention/procedure/surgery"
  To gather information, a questionnaire consisting of two sections, the first section, demographic characteristics including age, and weight, and the second section consisting analgesia scale was used.This tool assesses pain in pediatric patients, preverbal children, and those who cannot express their pain verbally or accurately and is dependent on the assessment by the researcher based on the criteria of this scale. In this project, zero is analgesia, 1-3 is for mild pain, 4-6 is for moderate pain, and 7-10 is for severe pain the Face Legs a useful tool for parents to detect pain in their infants and young children. and toddlers

SECONDARY OUTCOMES:
Differences between children pain scale after 6h | Differences between children who underwent circumcision' surgery with or without caudal block anesthesia in the average pain scores at the various time points, postoperative analgesia between children pain scores after 6hours
  Face, Legs, Activity, Cry, Consolability (FLACC) analgesia scale was used . The scores were observed and recorded during the first 5 min post op then 20 min, 30 min, and 60 min in Post Anesthesia Care unit. this scale is a standard tool to measure pain severity in which pain severity is scored from zero (analgesia) to 10 (maximum pain). This tool assesses pain in pediatric patients, preverbal children, and those who cannot express their pain verbally or accurately and is dependent on the assessment by the researcher based on the criteria of this scale. In this project, zero is analgesia, 1-3 is for mild pain, 4-6 is for moderate pain, and 7-10 is for severe pain .the pain scores were recorded at the various time points, postoperative analgesia between children pain scores after 6hours

CONTACTS AND LOCATIONS:
Overall Officials: Rashed A Albanna, consultant, Study Director — salmanyia medical complex
Locations (1):
- Salmanyia Medical Complex, Manama, Bahrain

IPD SHARING:
Plan to Share IPD: Yes
CONSORT checklist was used for the enrolment and allocation of patients, Children undergoing circumcision surgery under General Anesthesia (GA) with CB Group A and DPNB Group B, and systemic opioid Group C.
  inclusion and exclusion standards: After obtaining approval from the research approval serial number institution Review Board IRB number 7 0130623, informed written consent was obtained from the parents of 90 boys (ASA physical status I), aged from three months up to three years scheduled to undergo circumcision surgery,
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data is ready to upload starting 1/5/2023 end 20\8\2023
Access Criteria: All 90 patients poysAll statistical work will be carried out using Spss version 27 (Spss Inc., Chicago, USA) and Prism GraphPad version 9.4.1 (GraphPad, San Diego, USA) The categorical and numerical variables and demographic data of three groups were collected and reviewed by two authors.

REFERENCES:
- [Background] Gawe ZA, Isa HM, Almashaur MM, Haider F, Almulla K. The Effect of Caudal Anesthesia Block on Perioperative Pain Control and Reduction of the Anesthetic Agent in Pediatric Infraumbilical Surgery: A Prospective Randomized Trial Study. Anesth Essays Res. 2022 Jul-Sep;16(3):301-306. doi: 10.4103/aer.aer_64_22. Epub 2022 Nov 2. PMID 36620118
- [Background] Sandeman DJ, Reiner D, Dilley AV, Bennett MH, Kelly KJ. A retrospective audit of three different regional anaesthetic techniques for circumcision in children. Anaesth Intensive Care. 2010 May;38(3):519-24. doi: 10.1177/0310057X1003800317. PMID 20514962
- [Background] Metzelder ML, Kuebler JF, Glueer S, Suempelmann R, Ure BM, Petersen C. Penile block is associated with less urinary retention than caudal anesthesia in distal hypospadia repair in children. World J Urol. 2010 Feb;28(1):87-91. doi: 10.1007/s00345-009-0420-2. Epub 2009 May 23. PMID 19466428
- [Result] Cyna AM, Middleton P. Caudal epidural block versus other methods of postoperative pain relief for circumcision in boys. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD003005. doi: 10.1002/14651858.CD003005.pub2. PMID 18843636
- [Result] Ekstein M, Weinbroum AA, Ben-Chaim J, Amar E, Schvartz R, Klein Y, Bar-Yosef Y. Comparison of Caudal Block vs. Penile Block vs. Intravenous Fentanyl Only in Children Undergoing Penile Surgery: A Prospective, Randomized, Double Blind Study. Front Pediatr. 2021 Mar 26;9:654015. doi: 10.3389/fped.2021.654015. eCollection 2021. PMID 33842412
- [Result] Walker BJ, Long JB, Sathyamoorthy M, Birstler J, Wolf C, Bosenberg AT, Flack SH, Krane EJ, Sethna NF, Suresh S, Taenzer AH, Polaner DM, Martin L, Anderson C, Sunder R, Adams T, Martin L, Pankovich M, Sawardekar A, Birmingham P, Marcelino R, Ramarmurthi RJ, Szmuk P, Ungar GK, Lozano S, Boretsky K, Jain R, Matuszczak M, Petersen TR, Dillow J, Power R, Nguyen K, Lee BH, Chan L, Pineda J, Hutchins J, Mendoza K, Spisak K, Shah A, DelPizzo K, Dong N, Yalamanchili V, Venable C, Williams CA, Chaudahari R, Ohkawa S, Usljebrka H, Bhalla T, Vanzillotta PP, Apiliogullari S, Franklin AD, Ando A, Pestieau SR, Wright C, Rosenbloom J, Anderson T; Pediatric Regional Anesthesia Network Investigators. Complications in Pediatric Regional Anesthesia: An Analysis of More than 100,000 Blocks from the Pediatric Regional Anesthesia Network. Anesthesiology. 2018 Oct;129(4):721-732. doi: 10.1097/ALN.0000000000002372. PMID 30074928
- [Result] Baird R, Guilbault MP, Tessier R, Ansermino JM. A systematic review and meta-analysis of caudal blockade versus alternative analgesic strategies for pediatric inguinal hernia repair. J Pediatr Surg. 2013 May;48(5):1077-85. doi: 10.1016/j.jpedsurg.2013.02.030. PMID 23701786
- [Result] H G Salama, M H Elsersi, T S Shabana, J M Mahanna caudal block versus penile block for postoperative analgesia in children undergoing hypospadias repair, QJM: An International Journal of Medicine, Volume 113, Issue Supplement_1, March 2020, hcaa052.006
- Available data/document: Individual Participant Data Set: 70130623 — https://www.moh.gov.bh/Contact/SMC — This study was ethically approved by the Research and Research Ethics Committee Government Hospitals, Salmaniya Medical Complex (SMC), Kingdom of Bahrain, institution review board, (IRB) approval number: 70130623, which includes the use of patient data for research and educational purposes was obtained from all the patients/control's parents/guardians before the intervention. This study followed the guidelines laid down in the Declaration of Helsinki of 1975, and as revised in Edinburgh 2000.

DOCUMENTS (3):
  • Study Protocol (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT06086106/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT06086106/SAP_001.pdf
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT06086106/ICF_002.pdf